CLINICAL TRIAL: NCT06681012
Title: Gelsectan® in the Treatment of Patients With Diarrhoea-predominant Irritable Bowel Syndrome: a Multicentre, Randomized, Double-blind, Parallel-group, Placebo-controlled Study
Brief Title: Gelsectan® in the Treatment of Patients With Diarrhoea-predominant Irritable Bowel Syndrome
Acronym: GIANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Devintec Sagl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DVT2024
Record Dates: First submitted 2024-10-25; First posted 2024-11-08 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Syndrome (IBS); Irritable Bowel Syndrome of Diarrhea Type (IBS-D)
Keywords: Gelsectan; Irritable Bowel Syndrome (IBS); Irritable Bowel Syndrome of Diarrhea type (IBS-D)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gelsectan® (Experimental): Gelsectan® is a class III CE-marked medical device under the Regulation (EU) 2017/745 (MDR), which has been present on the EU market since 2017. Gelsectan® medical device consists of non-sterile capsules containing film-forming compounds (Xyloglucan, Pea protein, grape seed extract, and Xylo-oligosaccharide) indicated for symptomatic relief and prevention of IBS symptoms.
  Interventions: Device: Gelsectan®
- Placebo (Placebo Comparator): Placebo capsule, comparable in size, appearance and taste, packaging and labelling, as well as mode and schedule of administration to the IMD (i.e., Gelsectan®).
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: Gelsectan® — Oral capsules are to be taken twice a day for 2 months (two capsules in the morning before breakfast and two capsules in the evening before dinner during the first 4 weeks of treatment; one capsule in the morning and one in the evening during the following 4 weeks of treatment).
  Arms: Gelsectan®
Drug: Placebo — Oral capsules are to be taken twice a day for 2 months (two capsules in the morning before breakfast and two capsules in the evening before dinner during the first 4 weeks of treatment; one capsule in the morning and one in the evening during the following 4 weeks of treatment).
  Arms: Placebo

SUMMARY:
Irritable Bowel Syndrome (IBS) is one of the major Disorders of Gut-Brain Interaction (DGBI) and the most frequent reasons for referral to both primary care providers and gastroenterologists.IBS is not a life-threatening disease, but imposes a significant burden on society, entailing a decrease in patients' Quality of Life (QoL), elevated rates of psychological comorbidities and loss of work productivity, which might be the greatest in subjects with IBS-D, for whom the fear of incontinence in a social situation can be especially debilitating. Moreover, IBS is associated with significant direct and indirect healthcare costs and has a considerable socioeconomic impact on society.

Treatment strategy for IBS is usually based on predominant symptoms and their severity, and requires a strong patient-physician relationship, as well as both non-pharmacological and pharmacological approaches. Lifestyle interventions, such as dietary modifications, physical activity and lifestyle adjustments, and stress reduction/psychological therapy represent the most important initial non-pharmacological clinical approach for IBS patients, especially for those with mild disease. First-line pharmacological options for IBS-D include antidiarrheals, mainly loperamide, to control diarrhoea, as well as antispasmodic drugs to relieve IBS symptoms, in particular abdominal pain. Second-line therapies indicated for the treatment of global IBS-D symptoms include rifaximin, 5-Hydroxytryptamine (5-HT)3 receptor antagonists (alosetron, ondansetron and ramosetron) and eluxadoline. Other treatments recommended in patients with IBS-D consist of Tricyclic Anti-Depressants (TCAs) and bile acid sequestrants.

Notably, management of patients with IBS is challenging since diagnosis and treatment could require several therapeutical strategies with often partial and unsatisfactory results. Indeed, most patients with IBS are dissatisfied with their current therapy and 34% report no symptom control, according to the IBS Global Impact Report of 2018.

At present, there is a growing interest in therapeutic approaches for IBS-D aimed at improving intestinal barrier integrity for a more efficient control of symptoms, considering that an intestinal epithelial barrier dysfunction and mucosal immune activation have been suggested as a central mechanism in IBS-D pathophysiology. In this perspective, film-forming agents capable of protecting the intestinal mucosal barrier, such as Xyloglucan (XG) and Pea protein may represent a valid alternative therapeutic option for the management of IBS-D.

Gelsectan® is a CE-marked medical device under the European Union (EU) Medical Device Regulation (MDR) 2017/745, whose classification under the MDR is class III. Gelsectan® contains XG, Pea protein, grape seed extract, and Xylo-Oligosaccharides (XOS) and is indicated for symptomatic relief and prevention of chronic or relapsing diarrhoea, abdominal tension, pain, bloating and flatulence, as well as protection and restoration of intestinal mucosal function. Based on previous non-clinical studies and two clinical investigations, Gelsectan® seems to be safe and exert a protective action on the intestinal mucosa, mediating the restoration of intestinal permeability and the improvement of gastrointestinal symptoms associated with IBS-D. In particular, a 28-day treatment with Gelsectan® significantly reduced IBS-D-associated diarrhoea, abdominal pain and bloating, with no related adverse events in a randomized, placebo-controlled, cross-over clinical study. Moreover, Gelsectan® treatment for 6 months was generally safe and effective in improving IBS severity, diarrhoea and bowel habit, as well as pain and bloating, in a recent multicentre, open-label, prospective, observational study. Of note, Gelsectan® was also mentioned in the recent clinical practice guidelines on IBS-D and functional diarrhoea of the United European Gastroenterology (UEG) and the European Society for Neurogastroenterology and Motility (ESNM), and a recent consensus on IBS conducted by a panel of Belgian gastroenterologists.

With these premises, the present study aims to further assess the performance and safety of Gelsectan® within the scope of its intended purpose, compared with placebo, on overall abdominal pain and symptoms in patients with IBS-D in a randomized, double-blind, parallel-group clinical study.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, age ≥18 years and ≤ 65 years.
2. Positive diagnosis of IBS, according to Rome IV diagnostic criteria, namely recurrent abdominal pain, on average, at least 1 day/week in the last 3 months associated with two or more of the following criteria:

   * related to defecation
   * associated with a change in frequency stool
   * associated with a change in form (appearance) of stool The above criteria must be fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis.
3. Positive diagnosis of IBS-D subtype based on Rome IV diagnostic criteria, i.e., more than 25% of bowel movements with a consistency of type 6 or type 7 (loose or watery stools) on the BSFS, and less than 25% of bowel movements with BSFS types 1 or 2 (hard or lumpy stools), on days with at least one abnormal bowel movement.
4. Negative results to any relevant additional tests or exams whenever deemed appropriate by the Investigator to exclude other disorders or causes of IBS symptoms.
5. At least one type 6 or type 7 bowel movement based on the BSFS on at least 4 days within the last week prior to randomization.
6. Weekly average score of 24-hours worst abdominal pain score ≥ 3 on NRS-11 in the last week prior to randomization.
7. Electronic diary (e-diary) completed on at least 11 of 14 days (≥ 75%) during the screening period (i.e., 2 weeks prior to randomization).
8. Willingness and capability to fulfil all tasks foreseen by the Clinical Investigation Plan (CIP).
9. Signed written informed consent.
10. Females of childbearing potential must have a negative urine pregnancy test (dipstick) at randomization and currently use or agree to use consistently and correctly (i.e., perfect use) a highly effective or acceptable effective contraceptive method for the individual subject and her partner(s) throughout the study treatment period and for at least one full contraceptive cycle (when applicable).

Exclusion criteria:

1. Presence of any relevant organic, systemic or metabolic disease (particularly significant history of cardiovascular, renal, neurological, endocrine, metabolic or hepatic disease) that would preclude participation in this study in the opinion of the Investigator, or abnormal laboratory values that will be deemed clinically significant on the basis of predefined values.
2. Known perforation and/or gastrointestinal obstruction.
3. Ascertained organic gastrointestinal diseases, including celiac disease, bile acid malabsorption or inflammatory bowel diseases (Crohn's disease, ulcerative colitis, diverticular disease, infectious colitis, ischemic colitis, microscopic colitis).
4. Presence of other intestinal motility disorders, such as biliary dyskinesia, gastroparesis, intestinal pseudo-obstruction, and narcotic bowel syndrome.
5. Previous major abdominal surgery (uncomplicated appendectomy, cholecystectomy, polypectomy, inguinal hernia surgery, or caesarean section are allowed unless within six months prior to screening).
6. Active malignancy of any type (except for non-invasive basal or squamous cell carcinoma of the skin), or history of a malignancy other than non-invasive basal or squamous cell carcinoma of the skin. Patients with a history of malignancies that have been surgically removed with no evidence of recurrence for at least five years and no treatment prior to screening are allowed to participate in the study.
7. History of allergy or hypersensitivity to any of the investigational product ingredients or excipients.
8. Current use of Gelsectan®.
9. Use of loperamide or antispasmodics (i.e., direct smooth muscle relaxants, anticholinergic agents and calcium channel blockers) in the 14 days prior to randomization.
10. Concomitant use (starting from screening) of weak and potent opioids, 5-HT3 antagonists, such as alosetron and ondansetron, bile acid sequestrants, eluxadoline or any other drug/supplement known to significantly interfere with abdominal pain, stool frequency and consistency and/or intestinal permeability (except for those allowed as rescue therapy starting from randomization), including but not limited to corticosteroids, aminosalicylates, immunosuppressants and biologicals.
11. Prior and concomitant use of probiotics/prebiotics/synbiotics or rifaximin starting from 28 days prior to randomization. Other oral antibiotics and topical antibiotics are allowed.
12. Any major psychiatric unstable disorder, including eating disorders, and use of antidepressant or anxiolytic agents, unless used at a stable dose for at least 6 weeks prior to randomization.
13. History or current evidence of laxative abuse within 5 years prior to screening.
14. Recent history (within 12 months prior to screening) or suspicion of alcohol abuse or drug addiction.
15. Treatment with any investigational drug or medical device within 30 days prior to randomization, or current participation in other clinical trials or investigations.
16. Pregnancy or breastfeeding or intention to look for pregnancy throughout the whole study duration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Effect of Gelsectan® on the composite response rate for abdominal pain and stool consistency over the 8-week treatment period, at the end of treatment, in patients with IBS-D, according to Rome IV criteria. | From enrollment to the end of treatment at 8 weeks
  Proportion of composite responders over 8 weeks determined at the End of Treatment.
  A composite responder is defined as a patient who meet the following criteria for at least 50% of the 8-week treatment period:
  * Pain response criteria: reduction of at least 30% in the weekly average score of the 24-hour worst abdominal pain compared with baseline, measured with the 11-point Numeric Rating Scale (from 0=none to 10=worst possible pain) AND
  * Stool consistency response criteria: reduction of at least 50% in the number of days per week with at least one stool that has a consistency of BSFS types 6 or 7 compared with baseline, measured daily using the Bristol Stool Form Scale - BSFS (from 1=separate hard lumps, like nuts to 7=watery, no solid pieces).
  A patient needs to fulfil both aforementioned response criteria for abdominal pain and stool consistency in the same week to be considered a responder for that week.

SECONDARY OUTCOMES:
Effect of Gelsectan® on overall IBS-D symptoms: composite response rate for abdominal pain and stool consistency over 4-week intervals | From enrollment to the end of treatment at 8 weeks and each 4-week interval, as well as the 4-week post-treatment period
  Proportion of composite responders over each 4-week intervals.
  A composite responder is defined as a patient who meet the following criteria for at least 50% of the 8-week treatment period:
  * Pain response criteria: reduction of at least 30% in the weekly average score of the 24-hour worst abdominal pain compared with baseline, measured with the 11-point Numeric Rating Scale (from 0=none to 10=worst possible pain) AND
  * Stool consistency response criteria: reduction of at least 50% in the number of days per week with at least one stool that has a consistency of BSFS types 6 or 7 compared with baseline, measured daily using the Bristol Stool Form Scale - BSFS (from 1=separate hard lumps, like nuts to 7=watery, no solid pieces).
  A patient needs to fulfil both aforementioned response criteria for abdominal pain and stool consistency in the same week to be considered a responder for that week.
Effect of Gelsectan® on overall IBS-D symptoms: Proportion of pain responders | From enrollment to the end of treatment at 8 weeks and each 4-week interval, as well as the 4-week post-treatment period
  Proportion of pain responders, defined as patients who meet the pain response criteria (i.e., reduction of at least 30% in the weekly average score of the 24-hour worst abdominal pain compared with baseline) for at least 50% of the observation period.
  The standard 11-point Numeric Rating Scale (NRS-11) (from 0=none to 10=worst possible pain imaginable) will be used for the measure of pain.
Effect of Gelsectan® on overall IBS-D symptoms: Proportion of stool consistency responders | From enrollment to the end of treatment at 8 weeks and each 4-week interval, as well as the 4-week post-treatment period
  Proportion of stool consistency responders, defined as patients who meet the stool consistency response criteria (i.e., reduction of at least 50% in the number of days per week with at least one stool that has a consistency of BSFS types 6 or 7 compared with baseline) for at least 50% of the observation period.
  Stool consistency will be measured daily using the Bristol Stool Form Scale - BSFS (from 1=separate hard lumps, like nuts to 7=watery, no solid pieces).
Effect of Gelsectan® on overall IBS-D symptoms: Mean 24-hour worst abdominal pain score | From enrollment to the end of the 12 weeks study period
  Mean 24-hour worst abdominal pain score, as self-assessed by patients daily up to Week 12 using the Numeric Rating Scale (NRS-11) (from 0=none to 10=worst possible pain imaginable)
Effect of Gelsectan® on overall IBS-D symptoms: Mean stool type | From enrollment to the end of the 12 weeks study period
  Mean number of days/week with a BSFS type ≤ 2, ≥ 3 and ≤ 5, and ≥ 6, as well as changes from baseline, as self-assessed by patients daily up to Week 12 through the Bristol Stool Form Scale - BSFS (from 1=separate hard lumps, like nuts to 7=watery, no solid pieces).
Effect of Gelsectan® on overall IBS-D symptoms: Mean number of stools/day | From enrollment to the end of the 12 weeks study period
  Mean number of stools/day (average daily frequency of defecation)
Effect of Gelsectan® on overall IBS-D symptoms: Mean weekly average score for bloating | From enrollment to the end of the 12 weeks study period
  Mean weekly average score for bloating, as self-assessed by patients using a 7-point Likert scale (ranging from 0 to 6, where 0= not bad/bothersome at all and 6= extremely bad/bothersome)
Effect of Gelsectan® on overall IBS-D symptoms: Mean weekly average score for urgency of defecation | From enrollment to the end of the 12 weeks study period
  Mean weekly average score for urgency of defecation, as self-assessed by patients weekly using a 7-point Likert scale (ranging from 0 to 6, where 0= no urgency at all and 6= a very great deal of urgency)
Effect of Gelsectan® on IBS symptom severity: Proportion of patients with global improvement of IBS | From enrollment to the end of treatment at 8 weeks and after 4-week post-treatment period
  Proportion of patients with global improvement of IBS, defined as a score of at least 4 on the IBS Global Assessment of Improvement (IBS-GAI).
  IBS-GAI score ranging from 0 to 6 (where 0 = "substantially worse", 1 = "moderately worse", 2 = "slightly worse", 3 = "unchanged", 4 = "slightly improved", 5 = "moderately improved", and 6 = "substantially improved").
Effect of Gelsectan® on IBS symptom severity measured by the IBS-Symptom Severity Scale score | From enrollment to the end of treatment at 8 weeks and after 4-week post-treatment period
  Change from baseline in IBS severity, as measured by the IBS-Symptom Severity Scale (IBS-SSS) score.
  IBS-SSS is a validated five-item questionnaire measuring the frequency and intensity of abdominal pain, the severity of abdominal distension, the dissatisfaction with bowel habits, and the interference of IBS with daily life. Each item is rated from 0 to 100, with a total score ranging from 0 to 500, with higher scores indicating a greater severity. Severity of IBS can be graded as mild (<175), moderate (175-300), or severe (>300) based on the IBS-SSS total score.
Effect of Gelsectan® on work productivity and activity impairment due to IBS | From enrollment to the end of the 12 weeks study period
  Change from baseline of work productivity and activity impairment due to IBS, as measured by the Work Productivity and Activity Impairment (WPAI):IBS questionnaire scores.
  WPAI:IBS is a validated questionnaire consisting of six items intended to assess work productivity and daily activity impairment due to IBS in the preceding 7 days (Visual Analogue Scale [VAS] from 0 to 10) and daily activity impairment resulting from IBS (VAS from 0 to 10).
  WPAI:IBS scores are represented as percentages (range of 0-100%), with higher percentages indicating a greater work productivity loss and daily activity impairment.
Effect of Gelsectan® on quality of life as measured by World Health Organization Quality of Life Brief Version (WHOQOL-BREF) | From enrollment to the end of the 12 weeks study period
  Change from baseline of patient QoL, as measured by World Health Organization Quality of Life Brief Version (WHOQOL-BREF).
  The WHOQOL-BREF questionnaire is a validated measurement of QoL consisting of an abbreviated, 26-item version of the 100-item WHOQOL-100 QoL measure. The WHOQOL-BREF addresses four QoL domains, i.e., physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items), with each item graded on a 5-point Likert scale. Each domain score is calculated by multiplying by a factor of four the mean of all item scores. Domain scores are then transformed to a 0-100 scale, with higher scores indicating a better QoL.
Effect of Gelsectan® on depression symptoms | From enrollment to the end of the 12 weeks study period
  Change from baseline of symptoms of depression, as measured by the Patient Health Questionnaire (PHQ)-9 score.
  PHQ-9 is a nine-item questionnaire assessing depression symptoms according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) in the past two weeks, with each item score ranging from 0 (not at all) to 3 (nearly every day). The PHQ-9 total score is representative of depression severity and ranges from 0 to 27, by which depression is defined as mild (5-9), moderate (10-14), moderate (15-19) or severe (more than 20).
Use of rescue therapy | From enrollment to the end of treatment at 8 weeks
  Use of rescue therapy (type and posology) during treatment
Healthcare utilization | From enrollment to the end of treatment at 8 weeks
  Incidence of visits to patient's General Practitioner (GP), Emergency Room (ER) visits and unplanned hospitalizations (with length of stay)
Safety: adverse events and device deficiencies | From enrollment to the end of treatment at 8 weeks
  Incidence and type of all adverse events and device deficiencies throughout the study
Safety: changes in systolic and diastolic Blood Pressure | From enrollment to the end of treatment at 8 weeks
  Changes in systolic and diastolic Blood Pressure (mmHG)
Safety: changes in Heart Rate | From enrollment to the end of treatment at 8 weeks
  Changes in Heart Rate (bpm)
Safety: Changes in Respiratory Rate | From enrollment to the end of treatment at 8 weeks
  Changes in Respiratory Rate (breaths per minute)
Safety: Changes in the concentration of Glucose, Blood Urea Nitrogen (BUN), bilirubin, creatinine | From enrollment to the end of treatment at 8 weeks
  Changes in the concentration of Glucose, Blood Urea Nitrogen (BUN), bilirubin, creatinine (mg/dl)
Safety: Changes in the concentration of Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase | From enrollment to the end of treatment at 8 weeks
  Changes in the concentration of Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase (U/L)
Safety: Changes in White Blood Cell count, Platelet count, Red Blood Cell count | From enrollment to the end of treatment at 8 weeks
  Changes in White Blood Cell count, Platelet count, Red Blood Cell count
Safety: Changes in haemoglobin concentration | From enrollment to the end of treatment at 8 weeks
  Changes in haemoglobin (g/dl) concentration
Safety: Changes in haematocrit | From enrollment to the end of treatment at 8 weeks
  Changes in haematocrit (%)
Safety: changes in urine specific gravity | From enrollment to the end of treatment at 8 weeks
  Changes in urine specific gravity
Safety: changes in urine pH | From enrollment to the end of treatment at 8 weeks
  Changes in urine pH
Safety: changes in urine protein, glucose, bilirubin, ketones, blood concentrations | From enrollment to the end of treatment at 8 weeks
  Changes in urine protein, glucose, bilirubin, ketones, blood concentrations (mg/dl)

OTHER OUTCOMES:
Intestinal permeability: percentage fractional excretion of lactulose, mannitol and sucralose after triple sugar test | From enrollment to the end of treatment at 8 weeks
  Changes in the percentage fractional excretion of lactulose, mannitol and sucralose after triple sugar (lactulose, mannitol and sucralose) test (patients' urine samples)
Intestinal permeability: Lactulose/Mannitol Ratio and Sucralose/Mannitol Ratio after triple sugar test | From enrollment to the end of treatment at 8 weeks
  Changes in Lactulose/Mannitol Ratio and Sucralose/Mannitol Ratio in urine samples measured by Gas Chromatography-Mass Spectrometry (GC-MS) after triple sugar (lactulose, mannitol and sucralose) test (patients' urine samples)

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (6):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola, Bologna, BO
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation, Milan
  - AOU Federico II di Napoli, Napoli
  - Azienda Ospedale Università Padova, Padua
  - Azienda Ospedaliero Universitaria Pisana (AOUP), Pisa
  - S. Andrea University Hospital, Roma
- Spain (2):
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No